CLINICAL TRIAL: NCT04809870
Title: Esophagectomy in Patients With Liver Cirrhosis - an Observational Study
Brief Title: Esophagectomy in Patients With Liver Cirrhosis
Status: Completed | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Other Study IDs: UKE Hamburg
Record Dates: First submitted 2021-03-18; First posted 2021-03-22 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Esophageal Cancer; Liver Cirrhosis
Keywords: esophagectomy
MeSH Terms: conditions — Esophageal Neoplasms; Liver Cirrhosis | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- LC (liver cirrhotic patients): Patients with concomitant liver cirrhosis
  Interventions: Procedure: surgery
- Non-LC (non liver cirrhotic patients): Patients without concomitant liver cirrhosis
  Interventions: Procedure: surgery

INTERVENTIONS:
Procedure: surgery — retrospective comparison of esophagectomy for esophageal cancer in patients with or without concomitant liver cirrhosis

SUMMARY:
Retrospective and confounder adjusted comparison of perioperative and longterm outcomes of patients requiring an esophagectomy for esophageal cancer with and without concomitant liver cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* primary esophageal cancer with indication for curative treatment
* follow up period ≥ 5 years
* LC cohort: pre- or intraoperative histological proof of liver cirrhosis

Exclusion Criteria:

* recurrent esophageal cancer
* missing indication for curative treatment of esophageal cancer
* esophagectomy for benign esophageal lesions

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: retrospective analysis of a prospective maintained database of EC patients operated at the institution between 2012 to 2016
Sampling Method: Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-03-18 (Actual); Study Completion 2021-04-10 (Actual)

PRIMARY OUTCOMES:
Long-term survival | 5 years

SECONDARY OUTCOMES:
Major complication | 90 days postoperatively
  Clavin Dindo ≥ 3
Anastomotic leakage rate | 90 days postoperatively
  Rate of endoscopically diagnosed anastomotic leakage
Sepsis rate | 90 days postoperatively
  Rate of participants with ≥ 2 points in Sepsis-related organ failure (SOFA) score within hospital stay
Renal failure rate | 90 days postoperatively
  Rate of acute kidney insufficiency (AKI) II-III (AKI Kidney Disease: Improving Global Outcomes (KDIGO) Guidelines)
Hepatic failure rate | 90 days postoperatively
  Number of participants with clinical diagnosis: coagulopathy, icterus and potentially hepatic encephalopathy
Cardiac complication | 90 days postoperatively
  cardiac complication requiring pharmacological treatment or intervention and / or ICU surveillance
Chylus fistula rate | 90 days postoperatively
  Concentration of triglycerides (TG) in drain fluids ≥ 3 times TGs i.s.
Pulmonary complications | 90 days postoperatively
  Pneumonia requiring antibiotics, ventilatory insufficiency requiring supportive therapy

CONTACTS AND LOCATIONS:
Overall Officials: Reeh, MD, Principal Investigator — 1Department of General, Visceral and Thoracic Surgery, University Hospital Hamburg-Eppendorf
Locations (1):
- University of Hamburg Medical Institutions, Hamburg, Germany